CLINICAL TRIAL: NCT01257282
Title: Prevalence and Prognostic Value of Unrecognised Myocardial Injury in Stable Coronary Artery Disease (PUMI)- a Multicenter, Observational Cohort Study.
Brief Title: Prevalence and Prognostic Value of Unrecognized Myocardial Injury in Stable Coronary Artery Disease (PUMI)
Acronym: PUMI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Uppsala University (Other)
Responsible Party: professor Bertil Lindahl, Uppsala Clinical Research Centre
Other Study IDs: U-07-001
Record Dates: First submitted 2010-12-06; First posted 2010-12-09 (Estimated); Last update posted 2010-12-09 (Estimated); Status verified 2010-12

CONDITIONS: Stable Angina Pectoris
MeSH Terms: conditions — Angina, Stable

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma samples for biochemical markers. Whole blood samples for extraction of DNA for genetic analysis.
Oversight: Data Monitoring Committee: No

SUMMARY:
This study includes patients with stable coronary artery disease without previously known myocardial infarction, and investigates the prevalence of clinically unrecognized myocardial damage and its prognostic implication.

DETAILED DESCRIPTION:
A substantial portion of all myocardial infarctions are not clinically recognized, but the myocardial damage can be recognized afterwards e g by magnetic resonance imaging (MRI). This study includes patients with stable coronary artery disease without previously known myocardial infarction, and investigates the prevalence of clinically unrecognised myocardial damage (UMI), and the prognostic value of UMI regarding new cardiac events.

In a subset of the patients, the biologic intra-individual variability of troponin and other biochemical markers will be investigated (substudy protocol).

ELIGIBILITY:
Inclusion Criteria:

* symptoms of stable angina pectoris according to the treating physician
* scheduled for coronary angiography
* written informed consent

Exclusion Criteria:

* pathological Q-wave in the 12-lead resting ECG
* known previous myocardial infarction
* previous PCI (percutaneous coronary intervention) or CABG (coronary artery bypass graft)
* history of congestive heart failure
* anything that contraindicates a MRI investigation (e.g. pacemaker, claustrophobia, intracranial clips)
* lack of suitability for participation in the trial, for any reason, as judged by the Investigator.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with stable coronary artery disease without previously known myocardial infarction or coronary intervention
Sampling Method: Non-Probability Sample
Enrollment: 275 (Estimated)
Dates: Start 2007-09; Primary Completion 2013-03 (Estimated); Study Completion 2013-03 (Estimated)

PRIMARY OUTCOMES:
Cardiac events defined as a composite of death, resuscitated cardiac arrest, spontaneous acute myocardial infarction and hospitalisation for congestive heart failure or unstable angina. | 24 months

SECONDARY OUTCOMES:
Presence of unrecognized myocardial infarction | Baseline
Size and localisation of unrecognized myocardial infarction | Baseline
Degree and localization of artherosclerotic lesions at a coronary angiogram | Baseline
Procedure related acute myocardial infarction | 5 years
Left ventricular mass and dimensions, levels of troponin and other biochemical markers, electrocardiography (ECG), anthropometric data | Baseline
Long-term mortality, cardiac mortality and incidence of acute myocardial infarction | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Bertil Lindahl, professor, Principal Investigator — Uppsala University
Locations (6):
- Sweden (6):
  - Falu Hospital, Falun
  - Gävle Hospital, Gävle
  - Linköping University Hospital, Linköping
  - Örebro University Hospital, Örebro
  - Danderyds Hospital, Stockholm
  - Uppsala University Hospital, Uppsala

REFERENCES:
- [Derived] Nordenskjold AM, Hammar P, Ahlstrom H, Bjerner T, Duvernoy O, Eggers KM, Frobert O, Hadziosmanovic N, Lindahl B. Unrecognized Myocardial Infarction Assessed by Cardiac Magnetic Resonance Imaging--Prognostic Implications. PLoS One. 2016 Feb 17;11(2):e0148803. doi: 10.1371/journal.pone.0148803. eCollection 2016. PMID 26885831
- [Derived] Nordenskjold AM, Hammar P, Ahlstrom H, Bjerner T, Duvernoy O, Eggers KM, Frobert O, Hadziosmanovic N, Lindahl B. Unrecognized myocardial infarctions detected by cardiac magnetic resonance imaging are associated with cardiac troponin I levels. Clin Chim Acta. 2016 Apr 1;455:189-94. doi: 10.1016/j.cca.2016.01.029. Epub 2016 Jan 29. PMID 26828531
- [Derived] Hammar P, Nordenskjold AM, Lindahl B, Duvernoy O, Ahlstrom H, Johansson L, Hadziosmanovic N, Bjerner T. Unrecognized myocardial infarctions assessed by cardiovascular magnetic resonance are associated with the severity of the stenosis in the supplying coronary artery. J Cardiovasc Magn Reson. 2015 Nov 19;17:98. doi: 10.1186/s12968-015-0202-5. PMID 26585508